CLINICAL TRIAL: NCT04459169
Title: Early Echographic Screening of Cardiac Amyloidosis Using Red Flag Signals
Brief Title: Cardiac Amyloidosis : Diagnostic Using Red Flag Signals
Acronym: TEAM Red Flags
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH2-22
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: diagnostic algorithm — Cardiac amyloidosis diagnosed according to Gillmore's algorithm

SUMMARY:
Cardiac amyloidosis is an increasingly contributor of degenerative cardiac diseases. However, its frequency remains underestimated, and diagnosis is often realized at late stages of the disease. A larger use of clinical and echographic Red Flag signals during routine echocardiographic examination may enhance the identification of early stage of the disease.

DETAILED DESCRIPTION:
The objective is to evaluate the clinical and epidemiological aspects of cardiac amyloidosis using a systematic screening of even moderate left ventricular hypertrophy, taking into account the presence of Red Flag signals. Red Flag Signals will include history or symptoms of carpal tunnel syndrome, hearing loss, chronic gastrointestinal disorders, heart failure, cervical or lumbar stenosis, or echographic abnormalities such as apical sparring, increased left ventricular filling pressure, atrio-ventricular block.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of left ventricular hypertrophy defined by a parietal thickness (interventricular septum or posterior wall) ≥ 12 mm on the echocardiogram
2. Age equal or greater than 45 years
3. Current residency in Martinique, Guadeloupe or French Guyana
4. Ability to receive and understand research information
5. Ability to freely deliver informed written consent

Exclusion Criteria:

1. Pregnant or breastfeeding woman
2. Severe uncontrolled hypertension
3. Chronic hemodialysis
4. Person under legal protection measures (guardianship, curatorship, safeguard of justice), and person deprived of liberty

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caribbeans who the large share of populations from African origin may be associated with a high prevalence of Transthyretin amyloidosis.
  In this population, diagnosis procedure will be perform to any patient with Left Ventricular Hypertrophy (LVH) with wall thickness ≥ 12 mm associated with clinical manifestations (or Red Flag signals
Sampling Method: Probability Sample
Enrollment: 424 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of cardiac amyloidosis diagnosed according to Gillmore's algorithm | 3 months
  frequency of cardiac amyloidosis diagnosed according to Gillmore's algorithm at the end of the diagnosis procedures, using biological (presence of cell dyscrasia), imaging (myocardial staining of bone tracers), and tissue examination (Congo Red staining) variables

SECONDARY OUTCOMES:
Frequency genotype of Transthyretin cardiac amyloidosis according to Gillmore's algorithm | 5 months
  Evaluate the frequency of Transthyretin cardiac amyloidosis among subjects with even moderate left ventricular enlargement (wall thickness ≥ 12 mm), taking into account the presence or not of Red Flag signals
Distribution of Red Flag signals according to Transthyretin genotype | 5 months
  To Compare the distribution of Red Flag signals between wild type TTR cardiac amyloidosis and hereditary TTR cardiac amyloidosis
Diagnosis value of any Red Flag signal. | 5 months
  To evaluate the diagnostic performance of each of the Red Flag signals for the diagnosis of TTR cardiac amyloidosis
Elaboration of a pre-test probability score | 5 months
  To elaborate a pre-test probability score including the Red Flag signals, adapted to the Echo Lab settings.

CONTACTS AND LOCATIONS:
Overall Officials: Doctor INAMO Jocelyn, Study Director — CHU de Martinique
Locations (3):
- Centre Hospitalier de Basse-Terre, Basse-Terre, Guadeloupe
- Martinique (2):
  - CHU de Martinique, Fort-de-France
  - CHU de Martinique, La Trinité

REFERENCES:
- [Background] Benson MD, Waddington-Cruz M, Berk JL, Polydefkis M, Dyck PJ, Wang AK, Plante-Bordeneuve V, Barroso FA, Merlini G, Obici L, Scheinberg M, Brannagan TH 3rd, Litchy WJ, Whelan C, Drachman BM, Adams D, Heitner SB, Conceicao I, Schmidt HH, Vita G, Campistol JM, Gamez J, Gorevic PD, Gane E, Shah AM, Solomon SD, Monia BP, Hughes SG, Kwoh TJ, McEvoy BW, Jung SW, Baker BF, Ackermann EJ, Gertz MA, Coelho T. Inotersen Treatment for Patients with Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):22-31. doi: 10.1056/NEJMoa1716793. PMID 29972757
- [Background] Coelho T, Adams D, Silva A, Lozeron P, Hawkins PN, Mant T, Perez J, Chiesa J, Warrington S, Tranter E, Munisamy M, Falzone R, Harrop J, Cehelsky J, Bettencourt BR, Geissler M, Butler JS, Sehgal A, Meyers RE, Chen Q, Borland T, Hutabarat RM, Clausen VA, Alvarez R, Fitzgerald K, Gamba-Vitalo C, Nochur SV, Vaishnaw AK, Sah DW, Gollob JA, Suhr OB. Safety and efficacy of RNAi therapy for transthyretin amyloidosis. N Engl J Med. 2013 Aug 29;369(9):819-29. doi: 10.1056/NEJMoa1208760. PMID 23984729
- [Background] Di Nunzio D, Recupero A, de Gregorio C, Zito C, Carerj S, Di Bella G. Echocardiographic Findings in Cardiac Amyloidosis: Inside Two-Dimensional, Doppler, and Strain Imaging. Curr Cardiol Rep. 2019 Feb 12;21(2):7. doi: 10.1007/s11886-019-1094-z. PMID 30747298
- See also: Frequency of cardiac amyloidosis inpatients with unexplained left ventricular hypertrophy: The Caribbean Amyloidosis Study — https://www.em-consulte.com/article/1192918/article/frequency-of-cardiac-amyloidosis-inpatients-with-u